CLINICAL TRIAL: NCT04012502
Title: De-escalation of Chemoradiotherapy Density in HPV-related Oropharyngeal Carcinoma in Chinese Populations
Brief Title: De-escalation Protocols in HPV-related Oropharyngeal Carcinoma in Chinese Populations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chaosu Hu, Principal Investigator, Fudan University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019-OR001
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Oropharyngeal Carcinoma; De-escalation
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional treatment arm (Active Comparator): Two cycles docetaxel+cisplatin (TP) induction chemotherapy followed by concurrent cisplatin chemoradiotherapy with standard radiation dose (70Gy/35Fx) when responses to induction chemotherapy are less than 50% Partial Response(PR)
  Interventions: Other: conventional treatment
- Toxicities reduced treatment arm (Experimental): Two cycles docetaxel+cisplatin (TP) induction chemotherapy followed by reducing radiation dose(60Gy/30Fx) and omitting concurrent cisplatin chemotherapy when responses to induction chemotherapy are ≥ 50% Partial Response(PR)
  Interventions: Other: Toxicities reduced treatment

INTERVENTIONS:
Other: Toxicities reduced treatment — Two cycles docetaxel+cisplatin (TP) induction chemotherapy followed by reducing radiation dose(60Gy/30Fx) and omitting concurrent cisplatin chemotherapy when responses to induction chemotherapy are ≥ 50% Partial Response(PR)
  Arms: Toxicities reduced treatment arm
Other: conventional treatment — Two cycles docetaxel+cisplatin (TP) induction chemotherapy followed by concurrent cisplatin chemoradiotherapy with standard radiation dose (70Gy/35Fx) when responses to induction chemotherapy are less than 50% Partial Response(PR)
  Arms: conventional treatment arm

SUMMARY:
Human papillomavirus (HPV)-related oropharyngeal carcinoma are exquisitely radiosensitive. Several studies attempted to reduce the toxicities of treatments through reduced-dose radiation and showed promising results, but all data were collected from non-Chinese areas. Like nasopharyngeal carcinoma, oropharyngeal carcinoma may have different biological behavior and relationship with HPV infection. So the investigators studied whether toxicities reducing treatment with reduced radiation dose and omitted concurrent chemotherapy after good response to induction chemotherapy would maintain survival outcomes while improving tolerability for patients with HPV-positive oropharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of squamous cell carcinoma of oropharynx with IHC p16 positive or PCR HPV16 positive
* T1-2/N1-3M0（except T1N1M0 and single LN<3cm）or T3-4N0-3M0 according to UICC/AJCC 8th staging system
* Age ≥18
* No prior anti-tumor treatment
* Karnofsky Performance Score (KPS)≥70
* Adequate blood supply
* Informed consent obtained

Exclusion Criteria:

* cannot take contrast-MRI imaging
* Pregnant
* Combined with other malignant tumor (except basal cell carcinoma of skin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 year
  Progression Free Survival

SECONDARY OUTCOMES:
OS | 2 year
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Chaosu Hu, MD, Principal Investigator — Fudan University Shanghai cancer centre
Locations (1):
- Fudan Universtiy Shanghai Cancer Centre, Shanghai, Shanghai Municipality, China